CLINICAL TRIAL: NCT01821326
Title: Risk Factors for Rebleeding in Patients With Obscure Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Department of Gastroenterology,, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjyyxhk0831
Record Dates: First submitted 2013-03-23; First posted 2013-04-01 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Gastrointestinal Bleeding
Keywords: capsule endoscopy; obscure gastrointestinal bleeding; rebleeding; risk factors
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The investigators investigated the rebleeding rate the risk factors for rebleeding after long-term follow-up (≥12 months) in patients who underwent capsule endoscopy for obscure gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent capsule endoscopy in Shanghai Renji Hospital(China) from June 2002 to January 2012 for obscure gastrointestinal bleeding

Exclusion Criteria:

1. patients who did not undergo a gastroscopy and colonoscopy performed before capsule endoscopy examination; and
2. patients with follow-up examination for other know clinical diseases.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent CE in Shanghai Renji Hospital ( China )from June 2002 to January 2012 for OGIB
Sampling Method: Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2002-06; Primary Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, M.D. PhD., Principal Investigator — RenJi Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Obscure Gastrointestinal Bleeding
Started | 339
Completed | 339
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Obscure Gastrointestinal Bleeding
Number analyzed (Participants) | 339
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 200
  >=65 years | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (18.4)
Gender [Count of Participants; unit: Participants]
  Female | 162
  Male | 177
Region of Enrollment [Number; unit: participants]
  China | 339

OUTCOME MEASURES:

1. Primary Outcome: Rebleeding Rate
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Patients With Obscure Gastrointestinal Bleeding
Number analyzed (Participants) | 339
participants | 97

ADVERSE EVENTS:
Time Frame: 10 years
Arm/Group | Patients With Obscure Gastrointestinal Bleeding
Serious Adverse Events (participants affected / at risk) | 0/339
Other Adverse Events (participants affected / at risk) | 0/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Obscure Gastrointestinal Bleeding (N=339)
capsule endoscopy retention (Gastrointestinal disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No